CLINICAL TRIAL: NCT07334561
Title: Transcranial Electrical Stimulation for Comorbid Depression and Pain: From Technological Development to Clinical Translation in a Multicenter Trial
Brief Title: Multitarget Transcranial Direct Current Stimulation for Comorbid Depression and Chronic Pain: A Multicenter Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Shanghai 10th People's Hospital (Other); Shanghai Tongji Hospital, Tongji University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025-80
Record Dates: First submitted 2026-01-03; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Depression Disorder; Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- tDCS-DLPFC group (Active Comparator): They receive actual tDCS on purpose brain targets (DLPFC).
  Interventions: Device: tDCS
- Sham Group (Sham Comparator): They receive fake tDCS (no current) on purpose brain targets.
  Interventions: Device: tDCS
- tDCS-M1-DLPFC (Experimental): They receive actual tDCS on purpose brain targets (M1+DLPFC).
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — All the groups receive respective treatment 5 days/week for 2 weeks (10 sessions), with 2mA current, the anode on the F3 and C3, the cathode on the right supraorbital, 20min each session.
  Other Names: M1+DLPFC
  Arms: tDCS-M1-DLPFC
Device: tDCS — All the groups receive respective treatment 5 days/week for 2 weeks (10 sessions), with 2mA current only at the beginning and the end of the intervention for 30 seconds (0mA for 19min), the anode on the F3 and C3, the cathode on the right supraorbital, 20min each session.
  Other Names: sham tDCS
  Arms: Sham Group
Device: tDCS — All the groups receive respective treatment 5 days/week for 2 weeks (10 sessions), with 2mA current, the anode on the F3, the cathode on the right supraorbital, 20min each session.
  Other Names: DLPFC
  Arms: tDCS-DLPFC group

SUMMARY:
This clinical trial aims to investigate a novel non-pharmacological intervention, transcranial direct current stimulation (tDCS) for the treatment of comorbid depression and pain. The primary objectives are to optimize neurostimulation parameters through a multicenter randomized controlled design and to elucidate the underlying neural circuit-immune interaction mechanisms of this comorbidity. Participants with comorbid depression and chronic pain will be randomly assigned to receive active multi-target tES or sham stimulation. The intervention period will last for 2 weeks, followed by a series of post-treatment follow-up assessments. Researchers will compare the changes in depression severity (e.g., assessed by HAMD-24) and pain intensity (e.g., NRS, BPI) across groups to evaluate the efficacy. Secondary outcomes include pain perception, quuatitive sensory test, fMRI, MEG, metabolic markers, neurotransmitter and inflammation biomarkers. This study aims to provide a precise, individualized therapeutic strategy, reduce reliance on pharmacotherapy, and promote the development of domestic high-end medical devices.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-65 years;
2. Meet the diagnostic criteria for a depressive episode according to ICD-11, with current mild-to-moderate depressive symptoms (HAMD-24 score ≥8 and ≤34);
3. Report persistent pain lasting ≥3 months and score ≥4 on item 5 of the Brief Pain Inventory (BPI);
4. Maintain a stable anti-depression drug and psychological treatment plan (including dosage, drug type, or therapeutic approach) for at least four weeks prior to enrollment;
5. Right-handed, with normal hearing, vision, or corrected vision;
6. Able to voluntarily provide written informed consent to participate in the study and willing and capable of complying with all study procedures.

Exclusion Criteria:

1. Diagnosed with other psychiatric disorders, including schizophrenia spectrum disorders, bipolar I disorder (due to potential risk of manic episodes and contraindication of lithium or anticonvulsants), primary anxiety disorders, depression associated with severe somatic illness, etc.
2. Active suicidal ideation, defined as a score of 4 on item 3 of the HAMD-24.
3. Severe or treatment-resistant depression (HAMD-24 score ≥35, with current depressive episode lasting at least 2 years or failure to respond to two or more antidepressant treatments during the current episode).
4. Substance use disorder within the past 3 months.
5. Experience of malignant pain due to cancer pain syndrome, visceral pain (e.g., gastric pain), or referred pain (e.g., back pain from pancreatitis).
6. Neurological disorders associated with structural brain abnormalities (e.g., traumatic brain injury, recent stroke, brain tumor).
7. Having undergone neuromodulation treatments within the past 3 months, including electroconvulsive therapy (MECT), repetitive transcranial magnetic stimulation (rTMS), or transcranial electrical stimulation (tES).
8. Contraindications to transcranial electrical stimulation (e.g., intracranial metal implants, cardiac pacemaker, cochlear implant, skin lesions at stimulation sites, personal or family history of epilepsy).
9. Current or within the past 1 month use of medications affecting central nervous system excitability or pain, such as anticonvulsants, lithium, opioids, nonsteroidal anti-inflammatory drugs, and antipsychotics. Occasional as-needed use of acetaminophen as rescue medication is permitted but must be documented in detail in the study diary.
10. Signs of dementia or other severe cognitive impairment (MoCA score <17).
11. Severe or unstable somatic diseases, including but not limited to: neurological disorders (e.g., epilepsy, stroke, migraine, history of cranial surgery); cardiovascular diseases (e.g., uncontrolled hypertension, heart failure, arrhythmia, myocardial infarction); respiratory disorders (e.g., severe sleep apnea syndrome); malignancy or immunocompromised status; uncontrolled diabetes (fasting blood glucose >12 mmol/L).
12. Pregnancy or lactation.
13. Concurrent participation in another clinical trial, participation in any clinical trial within the past 90 days, or planned participation in another trial during the study period.
14. Any contraindications to magnetic resonance imaging (e.g., metal implants, claustrophobia, respiratory or motor impairments).
15. Inability to cooperate with study assessments.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
The reduction rate of the baseline BPI score at 1week, 2weeks, 6weeks | Baseline, 1week, 2weeks, 6weeks
  BPI score

SECONDARY OUTCOMES:
The reduction rate of the baseline HAMD score at 1week, 2weeks, 6weeks | Baseline, 1 week, 2 weeks, 6weeks
  HAMD score
Change from baseline QST at 2 weeks | Baseline, 2weeks
  Quantitative sensory test (heat/cold/press pain)
The reduction rate of the baseline PCS score at 1week, 2weeks, 6weeks | Bseline, 1week, 2weeks, 6weeks,
  Pain Catastrophizing Questionnaire
The reduction rate of the baseline GAD-7 score at 1week, 2weeks, 6weeks | Baseline, 1week, 2weeks, 6weeks
  Generalized Anxiety Disorder Scale -7
Change from Baseline CGI at 1 week, 2 weeks, 6 weeks | Baseline, 1 week, 2 weeks, 6 weeks
  Clinical Global Impression
Change from baseline Blood BDNF at 2 weeks, 6weeks | Baseline, 2 weeks, 6weeks
  BDNF in ng/mL
Change from baseline Blood inflammatory factors at 2 weeks, 6weeks | Baseline, 2 weeks, 6weeks
  Inflammatory factors (IL-1β, IL-6, TNF-α, CRP, IL-2, IL-10, TGF-β) in ng/mL
Change from baseline Blood lipid at 2 weeks, 6weeks | Baseline, 2 weeks, 6weeks
  Blood lipid (Triglyceride, Total Cholesterol, Low-density Lipoprotein, High-density Lipoprotein) in mmol/L
Change from baseline Blood Glucose at 2 weeks, 6 weeks | Baseline, 2 weeks, 6 weeks
  Blood Glucose in mmol/L
Change from baseline fNIRS at 2 weeks | Baseline, 2 weeks
  Near-infrared brain function detection
Change from baseline fMRI at 2 weeks | Baseline, 2 weeks
  Functional magnetic resonance imaging

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Shanghai Mental Health Center, Shanghai, Shanghai Municipality
  - Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Yes